CLINICAL TRIAL: NCT05612243
Title: Investigation of the Bioactivity of Yogurt Enriched With Probiotics and Polyphenols, Through Its Postprandial Effect on Specific Blood Biomarkers in Healthy Participants
Brief Title: Effect of Consumption of a Novel Functional Yogurt on Blood Biomarkers of Healthy Participants
Acronym: FB-CL1
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: ANTONIOS KOUTELIDAKIS (Other)
Collaborators: Democritus University of Thrace (Other); University of Ioannina (Other)
Responsible Party: Sponsor-Investigator, ANTONIOS KOUTELIDAKIS, Assistant Professor, University of the Aegean
Organization: University of the Aegean (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Health Services Research
Other Study IDs: 5047291
Record Dates: First submitted 2022-11-03; First posted 2022-11-10 (Actual); Last update posted 2022-12-06 (Actual); Status verified 2022-12

CONDITIONS: Healthy
Keywords: probiotics; antioxidants; blood biomarkers; functional yogurt; postprandial effect; polyphenols
MeSH Terms: interventions — Polyphenols

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Yogurt enriched with probiotics and polyphenols (Experimental): Participants will consume a meal including 200g of yogurt containing Lacticaseibacillus rhamnosus probiotics (3*10^9 cfu/g) immobilized on oat flakes (1g) and polyphenol-rich lyophilized extract (250mg) of Cistus Albidus (77,3 mg GAE/g), as well as two slices of white bread (80g) with butter (30g)
  Interventions: Other: Consumption of a meal with yogurt enriched with probiotics immobilized on oat flakes and polyphenols
- Yogurt enriched with probiotics (Active Comparator): Participants will consume a meal including 200g of yogurt containing Lacticaseibacillus rhamnosus probiotics (3*10^9 cfu/g) immobilized on oat flakes (1g), as well as two slices of white bread (80g) with butter (30g)
  Interventions: Other: Consumption of a meal with yogurt enriched with probiotics immobilized on oat flakes
- Plain yogurt with oat flakes (Placebo Comparator): Participants will consume a meal including 200g of plain yogurt containing oat flakes (1g), as well as two slices of white bread (80g) with butter (30g)
  Interventions: Other: Consumption of a meal with plain Yogurt with oat flakes

INTERVENTIONS:
Other: Consumption of a meal with yogurt enriched with probiotics immobilized on oat flakes and polyphenols — Participants will consume a meal including 200g of yogurt enriched with Lacticaseibacillus rhamnosus probiotics (3*10^9 cfu/g) immobilized on oat flakes (1g) and polyphenol-rich lyophilized extract (250mg) of Cistus Albidus (77,3 mg GAE/g), as well as two slices of white bread (80g) with butter (30g). Then blood biomarkers will be examined to determine the effect of functional yogurt on postprandial glycemia and lipemia
  Arms: Yogurt enriched with probiotics and polyphenols
Other: Consumption of a meal with yogurt enriched with probiotics immobilized on oat flakes — Participants will consume a meal including 200g of yogurt with Lacticaseibacillus rhamnosus probiotics (3*10^9 cfu/g) immobilized on oat flakes (1g), as well as two slices of white bread (80g) with butter (30g). Then blood biomarkers will be examined to determine the effect of probiotic-enriched yogurt on postprandial glycemia and lipemia.
  Arms: Yogurt enriched with probiotics
Other: Consumption of a meal with plain Yogurt with oat flakes — Participants will consume a meal including 200g of plain yogurt containing 1g of oat flakes, as a placebo, as well as two slices of white bread (80g) with butter (30g). Then blood biomarkers will be examined to determine the effect of probiotic-enriched yogurt on postprandial glycemia and lipemia.
  Arms: Plain yogurt with oat flakes

SUMMARY:
The purpose of the study is to assess the effect of a dietary intervention that includes the consumption of a novel functional yogurt (enriched with probiotics and polyphenols) on the blood biomarkers of healthy participants.

DETAILED DESCRIPTION:
After having been informed about the study and the potential risks, all participants giving written informed consent will undergo screening to determine eligibility for study entry (inclusion criteria). At baseline (t0), a fasting blood sample will be taken by venipuncture from the participants, and they will be randomly assigned in a double-blind manner (investigator and participant) to one of the intervention groups, i.e. meal including the consumption of the functional yogurt (yogurt enriched with probiotics and polyphenols) or consumption of yogurt enriched with probiotics or consumption of placebo yogurt. The participants have to finish their meals within 15 minutes (t1) and after the meal, blood sampling will be repeated for the times, t2 = 30 min, t3 = 90 min, t4 = 180min. After a washout period of 7 days, the participants will consume the functional yogurt, or the yogurt enriched with probiotics, or the placebo yogurt, in a cross-over design, and the blood sampling will be carried out as described above. Finally, after a washout period of 7 days, the participants will consume the functional yogurt, or the yogurt enriched with probiotics or the placebo yogurt in a cross-over design, and the blood sampling will be carried out as described above. Throughout the interventional period participants' dietary intake, anthropometrical data, medical history, and dietary habits will be monitored.

ELIGIBILITY:
Inclusion Criteria:

-healthy individuals aged 18-65 years old, of both sexes/genders

Exclusion Criteria:

* BMI > 30 kg/m^2
* contraceptive pills taking
* lactose intolerance or food allergy to any of the ingredients of the food under study
* probiotic supplements or medications that affect bowel function
* pregnant or lactating women
* illicit drug use or chronic alcoholism or total daily alcohol intake > 50 g/d
* people with a chronic condition (cancer, active liver disease, severe kidney dysfunction, severe stroke in the last six months and conditions associated with an increased risk of bleeding) or individuals with any other serious medical condition that may affect their ability to participate in a dietary intervention study
* individuals who are considered unreliable by the researcher or who have a shorter life expectancy than the expected duration of the study, due to some illness or if they are in any condition which in the researcher's opinion does not allow their safe participation in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2022-10-17 (Actual); Primary Completion 2022-12-10 (Estimated); Study Completion 2022-12-16 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in metabolic health | 3 hours
  Blood samples will be obtained after an overnight, 12-h fasting and 30, 90 and 180 min after meal consumption. Blood serum analysis will include assessment of lipidemic profile [i.e. Total Cholesterol (TC), Low-Density Lipoprotein Cholesterol (LDL-C), High-Density Lipoprotein Cholesterol (HDL-C), Triglycerides (TG)], insulin, cortisol and uric acid.
Change from baseline in blood glucose | 3 hours
  Blood samples will be obtained after an overnight, 12-h fasting and 30, 90 and 180 min after meal consumption. Blood plasma analysis will include assessment of glucose metabolism [i.e. Fasting Blood Glucose (FBG)]
Change from baseline in C-reactive protein (CRP) | 3 hours
  Blood samples will be obtained after an overnight, 12-h fasting and 30, 90 and 180 min after meal consumption.
Change from baseline in Oxidative stress | 3 hours
  Blood samples will be obtained after an overnight, 12-h fasting and 30, 90 and 180 min after meal consumption and serum analysis will be conducted with a free radical analytical system

CONTACTS AND LOCATIONS:
Overall Officials: Antonios E. Koutelidakis, Study Director — University of the Aegean
Locations (1):
- University of the Aegean, Myrina, Greece

REFERENCES:
- [Background] Fidelix M, Milenkovic D, Sivieri K, Cesar T. Microbiota modulation and effects on metabolic biomarkers by orange juice: a controlled clinical trial. Food Funct. 2020 Feb 26;11(2):1599-1610. doi: 10.1039/c9fo02623a. PMID 32016250
- [Background] Annuzzi G, Bozzetto L, Costabile G, Giacco R, Mangione A, Anniballi G, Vitale M, Vetrani C, Cipriano P, Della Corte G, Pasanisi F, Riccardi G, Rivellese AA. Diets naturally rich in polyphenols improve fasting and postprandial dyslipidemia and reduce oxidative stress: a randomized controlled trial. Am J Clin Nutr. 2014 Mar;99(3):463-71. doi: 10.3945/ajcn.113.073445. Epub 2013 Dec 24. PMID 24368433
- [Background] Gomes APO, Ferreira MA, Camargo JM, Araujo MO, Mortoza AS, Mota JF, Coelho ASG, Capitani CD, Coltro WKT, Botelho PB. Organic beet leaves and stalk juice attenuates HDL-C reduction induced by high-fat meal in dyslipidemic patients: A pilot randomized controlled trial. Nutrition. 2019 Sep;65:68-73. doi: 10.1016/j.nut.2019.03.004. Epub 2019 Mar 16. PMID 31029925